CLINICAL TRIAL: NCT01706094
Title: Head Position in Stroke Trial
Acronym: HeadPoST-Pilot
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Clinica Alemana de Santiago (Other)
Collaborators: The George Institute (Other)
Responsible Party: Principal Investigator, Veronica Olavarria, MD, MSc, Clinica Alemana de Santiago
Allocation: Not Applicable | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: HeadPoST1
Record Dates: First submitted 2012-10-11; First posted 2012-10-15 (Estimated); Last update posted 2015-12-04 (Estimated); Status verified 2015-12

CONDITIONS: Ischemic Stroke
Keywords: stroke; head position
MeSH Terms: conditions — Ischemic Stroke; Stroke | interventions — Head-Down Tilt

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- lying flat head position (Experimental): positioning the head of the bed at zero degrees during the first 48 hours from admission of patients with acute ischemic stroke Active Comparator: upright position of the head of the bed during 48 hours from admission of patients with acute ischemic stroke
  Interventions: Other: Head Position

INTERVENTIONS:
Other: Head Position — Head position during the first 48 hours from admission of patients with acute ischemic stroke.
  This trial is organized as a cluster randomised trial to a policy of flat head position or upright head position. Clusters will be months, so that all patients admitted during a given month will be positioned either in the flat down head position (intervention) or upright head position (control). This will allow health teams to follow a monthly protocol without changing position between patients.

SUMMARY:
A simplest manner to augment cerebral blood flow to irrigate the ischemic penumbra in acute ischemic stroke could be to place the patient in a 'lying flat' rather than upright head position. Given uncertainty over the balance of potential modest benefits and risks, and variability regarding the ideal head position policy for patients with acute ischemic stroke around the world, reliable randomized evidence is required to standardize clinical practice.

The main objectives of this pilot phase clinical trial are to determine the feasibility, safety and potential efficacy of a large-scale cluster randomized clinical trial to assess whether a simple nursing care policy - 'lying flat head position' - provides beneficial effects as compared to the standard upright head position in patients with acute ischemic stroke. The main efficacy outcome of the pilot phase is demonstration of increased mean cerebral blood flow velocity in the flat down compared to the upright head position, as assessed by transcranial Doppler to the medial cerebral arteries of patients with anterior circulation infarction. Secondary efficacy objectives are to demonstrate that the flat down head position improves neurological status at 7 days and disability at 90 days.

DETAILED DESCRIPTION:
Background: Several lines of investigation indicate there to be potential beneficial effects of interventions that augment cerebral blood flow (CBF) to irrigate the ischemic penumbra in acute ischemic stroke. The simplest manner to do this is to place the patient in a 'lying flat' rather than upright head position. However, any potential benefits on the brain may be offset by an increased hazard of aspiration pneumonia or exacerbation of cardiac failure in vulnerable patients. Given uncertainty over the balance of potential modest benefits and risks, and variability regarding the ideal head position policy for patients with acute ischemic stroke around the world, reliable randomized evidence is required to standardize clinical practice.

Aims: The main objectives of this pilot phase clinical trial are to determine the feasibility, safety and potential efficacy of a large-scale cluster randomized clinical trial to assess whether a simple nursing care policy - 'lying flat head position' - provides beneficial effects as compared to the standard upright head position in patients with acute ischemic stroke. The main efficacy outcome of the pilot phase is demonstration of increased mean cerebral blood flow velocity (CBFV) in the lying flat head position compared to the upright head position, as assessed by transcranial Doppler (TCD) to the medial cerebral arteries of patients with anterior circulation infarction. Secondary efficacy objectives are to demonstrate that the lying flat head position improves neurological status at 7 days and disability at 90 days.

Methods: Inclusion criteria include consecutive adult patients with acute ischemic stroke within 12 hours of onset admitted to participating centers. A cluster (month) method of randomization to lying flat or upright head position for 48 hours, stratified by site The primary outcome is change in mean CBFV measured by TCD at 24 hours. Secondary outcomes include proportion of adverse events at 7 days, distribution of NIHSS at 7 days, and distribution of mRS disability scale scores at 90 days. Sample size is 46 clusters of 2 patients totaling approximately 92 patients to detect an increase of 8.31 (CI 95% 4.82-12.0) cm/sec in average CBFV from 30° to 0° head position. This sample size will also allow detection of that difference with 90% power at a 5% significance level, considering an ICC of 0.037.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 or more years old
* Patients with an acute stroke corresponding to anterior circulation, a CT scan ruling out intracranial hemorrhage, presenting within 12 hours from symptom onset
* NIHSS ≥1
* Susceptible to be tilted down to the flat position or to 30º of the head
* There is uncertainty about the benefit/harm of head position during a minimum of 24 hours.
* Informed consent given

Exclusion Criteria:

* Contraindications to a flat head position (active vomiting, pneumonia, uncontrolled heart failure)
* Concomitant medical illness that would interfere with outcome assessment and follow-up
* Planned decompressive craniectomy or carotid endarterectomy.
* Absence of sonographic temporal window

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 92 (Actual)
Dates: Start 2013-01; Primary Completion 2015-07 (Actual); Study Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
Increased mean cerebral blood flow velocity (CBFV) in the lying flat compared to the upright head position | 24 hours
  The main efficacy outcome of the pilot phase is demonstration of increased mean cerebral blood flow velocity (CBFV) in the lying flat head position compared to the upright head position, as assessed by transcranial Doppler (TCD) to the medial cerebral arteries of patients with anterior circulation infarction.

SECONDARY OUTCOMES:
proportion of Serious adverse events. | 7 days
  Assessments of Serious adverse events at 7 days comparing between the two head positioning groups.

OTHER OUTCOMES:
Functional outcomes | 7 days and 90 days
  Secondary efficacy outcome are to demonstrate that the lying flat head position improves neurological status at 7 days and disability at 90 days, measured by modified Rankin Scale, in person or by telephone.

CONTACTS AND LOCATIONS:
Overall Officials: Veronica V Olavarria, MD, Msc, Study Director — Clinica Alemana de Santiago, Chile.
Locations (3):
- Royal Prince Alfred Hospital, Sydney, New South Wales, Australia
- Chile (2):
  - Hospital regional Dr. Lautaro Navarro Avaria, Punta Arenas, Region de Magallanes
  - Clinica Alemana de Santiago, Santiago, Santiago Metropolitan

REFERENCES:
- [Derived] Olavarria VV, Lavados PM, Munoz-Venturelli P, Gonzalez F, Gaete J, Martins S, Arima H, Anderson CS, Brunser AM. Flat-head positioning increases cerebral blood flow in anterior circulation acute ischemic stroke. A cluster randomized phase IIb trial. Int J Stroke. 2018 Aug;13(6):600-611. doi: 10.1177/1747493017711943. Epub 2017 Jun 5. PMID 28581366
- [Derived] Olavarria VV, Arima H, Anderson CS, Brunser A, Munoz-Venturelli P, Billot L, Lavados PM; HEADPOST Pilot Investigators. Statistical analysis plan of the head position in acute ischemic stroke trial pilot (HEADPOST pilot). Int J Stroke. 2017 Feb;12(2):211-215. doi: 10.1177/1747493016674955. Epub 2016 Oct 14. PMID 27742914
- [Derived] Brunser AM, Munoz Venturelli P, Lavados PM, Gaete J, Martins S, Arima H, Anderson CS, Olavarria VV. Head position and cerebral blood flow in acute ischemic stroke patients: Protocol for the pilot phase, cluster randomized, Head Position in Acute Ischemic Stroke Trial (HeadPoST pilot). Int J Stroke. 2016 Feb;11(2):253-9. doi: 10.1177/1747493015620808. PMID 26783317